CLINICAL TRIAL: NCT04724200
Title: Optimising a Digital Diagnostic Pathway for Heart Failure in the Community
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: INGN20CA503
Record Dates: First submitted 2021-01-05; First posted 2021-01-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: echocardiogram; NTproBNP; digital diagnosis
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Referred from primary care for investigation of suspected heart failure: All patients recruited to the OPERA trial will have been referred from their primary care clinician for investigation of a suspected diagnosis of heart failure.
  Interventions: Diagnostic Test: Echocardiogram

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Echocardiography plays a crucial role in the diagnosis of HF; it is the standard of care imaging modality used to confirm the diagnosis, it permits real-time imaging of the heart and quantitative assessment of cardiac structure and function, crucial for diagnosis.

SUMMARY:
This is a prospective, observational study. The primary aim is to assess the diagnostic accuracy of Artificial Intelligence (AI) analysis of Point of Care (POC) handheld transthoracic echocardiogram images (POC handheld echocardiogram) compared to the current gold-standard of transthoracic echocardiogram images acquired and analysed by a British Society of Echocardiography (BSE) accredited operator, using a standard echocardiogram machine (standard TTE), for the diagnosis of Heart Failure with reduced Ejection Fraction (HFrEF), in patients referred from the community for investigation of suspected new Heart Failure (HF).

DETAILED DESCRIPTION:
1. Demonstrate that in comparison to using the current gold standard of BSE accredited operator echocardiography within a HFDP, using AI enhanced analysis of POC handheld echocardiography is accurate and safe. This has the potential to improve access to timelier echocardiography in order to achieve earlier HF diagnosis and treatment, which is known to delay/prevent progression to HF hospitalisation. It will also provide useful information regarding the future feasibility of using AI enhanced analysis of POC handheld echocardiography in the community, for investigation of people with suspected new HF.
2. Facilitate the digitisation of an NHS Heart Failure diagnostic service in order to standardise and improve the quality of data collection and clinical care provided within the service.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals referred from the community who are awaiting HF diagnostic investigations, including echocardiography, to investigate for a suspected new diagnosis of HF

Exclusion Criteria:

1. Individuals less than 18 years of age
2. Individuals who have had an interim echocardiogram for another clinical reason, whilst on the outpatient echocardiogram waiting list for investigation of HF
3. Individuals with a previous ICD-10 diagnosis of HF in any coding position
4. Inability of the participant, in the opinion of the investigators, to understand and/or comply with study procedures, or any conditions that, in the opinion of the investigators, may render the participant unable to understand, attend and/or undergo study visit investigations
5. Inability to read and understand the PIS (provided in English only), and understand the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 864 participants, who have been referred for echocardiography to investigate a suspected new diagnosis of HF, but who have not been able to undergo echocardiographic testing yet due to additional barriers and delays to access imposed by the COVID-19 pandemic, will be recruited from the HF diagnostic pathway waiting list in NHS Greater Glasgow and Clyde between 1st December 2020 and 31st March 2021.
  Study visits would normally be undertaken within NHS Greater Glasgow and Clyde hospitals. For public health physical distancing compliance reasons, study visits will take place in the NHS Louisa Jordan hospital (situated within the Scottish Exhibition and Conference Centre), temporarily converted for NHS clinical use to manage demand vs capacity issues during the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 867 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Negative and positive predictive value (NPV and PPV) | 1 day
  NPV and PPV describe the proportions of postive and negative results that are true results
False positive | 1 day
  A results that wrongly indicates heart failure is present in the OPERA patient
False negative | 1 day
  A result that wrongly indicates heart failure is not present in the OPERA patient
sensitivity | 1 day
  the ability of a diagnostics test to correctly identify those with heart failure
specificity | 1 day
  the ability of a diagnostic test to correctly identify those without heart failure
Area under curve | 1 day
  area under receiver operator curve comparison of the standard TTE Vs AI analysed POC echocardiogram for the diagnosis of HFrEF in people referred from the community for investigation of suspected new HF

CONTACTS AND LOCATIONS:
Overall Officials: Clare Murphy, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- NHS Louisa Jordan, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed